CLINICAL TRIAL: NCT02118259
Title: Impact of Multidisciplinary Review of Drug Prescriptions on Patient Safety in a Residence for Dependent Elderly
Acronym: Rev-EHPAD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: LOCAL/2013/GL-01; 2013-A01590-45 (Other: RCB number)
Record Dates: First submitted 2014-04-16; First posted 2014-04-21 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-04

CONDITIONS: Geriatrics; Residence for Dependent Elderly; Health Services for the Aged
Keywords: Multidisciplinary review of drug prescriptions; Adverse drug events geriatric risk score; Residence for dependent elderly
MeSH Terms: interventions — Controlled Before-After Studies

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- The study population (Other): See inclusion and exclusion criteria.
  Intervention: Before-after study
  Interventions: Other: Before-after study

INTERVENTIONS:
Other: Before-after study — The before-after study is composed of a first observational phase followed by a proactive phase, and then finally by a second observational phase.
  The first observational phase corresponds to retrospective data-collecting for the information necessary for calculating the baseline ADE geriatric risk score.
  The proactive phase corresponds to a multidisciplinary review of drug prescriptions (especially long-term drugs) for all included patients in the residence.
  During the second observational phase, the same data as in the first observational phase will be collected a second time.

SUMMARY:
The main objective of the study is to show that the multidisciplinary review of drug prescriptions changes the adverse drug event (ADE) geriatric risk score (according to Trivalle and Ducimetière 2013) for patients living in the Nîmes University Hospital Residence for Dependent Elderly.

DETAILED DESCRIPTION:
The secondary objectives of this study are to assess and compare the following criteria before and after multidisciplinary review of drug prescriptions for patients in the Nîmes University Hospital Residence for Dependent Elderly:

A. the number of patients with at least one potentially inappropriate drug prescribed

B. the number of hospitalizations

C. death rate

D. the number of falls per patient and the rate of fallers

E. qualitative criteria describing the drug review

F. associated care costs

ELIGIBILITY:
Inclusion Criteria:

* The patient (or his/her legal representative) must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* The patient is available for 6 months of follow-up
* The patient has resided at the Nîmes University Hospital Residence for Dependent Elderly for at least the past 6 months

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection
* The patient (or his/her legal representative) refuses to sign the consent
* It is impossible to correctly inform the patient (or his/her legal representative)
* The patient has resided at the Nîmes University Hospital Residence for Dependent Elderly for less than 6 months

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 49 (Actual)
Dates: Start 2014-05; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Adverse Drug Events Geriatric Risk Score | change from Baseline to 6 months
  according to Trivalle and Ducimetière 2013

SECONDARY OUTCOMES:
The number of patients taking at least 1 potentially inappropriate drug according to Laroche criteria | During the proactive phase. Day 0.
  Laroche et al 2007.
Number of hospitalizations in the public sector (higher level care) | first observational phase (month -6 to day 0)
Number of hospitalizations in the public sector (higher level care) | second observational phase (day 0 to month 6)
Days of hospitalization in the public sector (higher level care) | first observational phase (month -6 to day 0)
Days of hospitalization in the public sector (higher level care) | second observational phase (day 0 to month 6)
Mortality | first observational phase (month -6 to day 0)
Mortality | second observational phase (day 0 to month 6)
The number of falls per patient | first observational phase (month -6 to day 0)
The number of falls per patient | second observational phase (day 0 to month 6)
The percentage of patients who fell | first observational phase (month -6 to day 0)
The percentage of patients who fell | second observational phase (day 0 to month 6)
The Anatomical Therapeutic Chemical classification for each revised drug | during the proactive phase (day 0)
The type of errors detected during drug review | during the proactive phase (day 0)
  Contra-indication, dosing, route, etc
The type of modification suggested during drug review | during the proactive phase (day 0)
  discontinuation, addition, substitution...
The acceptation rate for modifications suggested during drug review | during the proactive phase (day 0)
Associated care costs (€) | first observational phase (month -6 to day 0)
Associated care costs (€) | second observational phase (day 0 to month 6)

CONTACTS AND LOCATIONS:
Overall Officials: Géraldine Leguelinel, Pharm-D, Study Director — Centre Hospitalier Universitaire de Nîmes
Locations (2):
- France (2):
  - CHRU de Nîmes - Centre de Gérontologie de Serre Cavalier, Nîmes
  - CHRU de Nîmes - Hôpital Universitaire Carémeau, Nîmes